CLINICAL TRIAL: NCT00003302
Title: Breast MRI Protocol
Brief Title: MRI to Detect Breast Tumors in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Diagnostic
Other Study IDs: CDR0000066242; UPCC-ACR-6883
Record Dates: First submitted 1999-11-01; First posted 2004-03-01 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Biopsy; Magnetic Resonance Imaging; Mammography

INTERVENTIONS:
Procedure: biopsy
Diagnostic Test: magnetic resonance imaging
Diagnostic Test: mammography

SUMMARY:
RATIONALE: New imaging procedures, such as MRI, may improve the ability to detect breast tumors.

PURPOSE: Diagnostic study to determine the value of MRI in detecting breast tumors in women who have had suspicious mammographic or clinical examinations.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the performance of breast magnetic resonance imaging (MRI) in conjunction with mammography for the detection and characterization of lesions in women with suspicious mammographic or clinical examinations. II. Assess the incremental value of breast MRI to determine the local extent of cancer in these patients. III. Assess the value of breast MRI to determine the prevalence and characteristics of incidental enhancing lesions in the remainder of the breast.

OUTLINE: This is a multicenter study. Patients undergo a high resolution 3D post contrast magnetic resonance imaging (MRI) scan. Patients with enhancing abnormalities undergo a dynamic scan no less than 18 hours later. Some patients may require a third scan if a core biopsy is to be performed. Patients who are ultimately found to have cancer are assessed for extent of cancer including measurement of the index lesion and identification of other present foci of cancer in relation to the index lesion. Further histological diagnosis of index lesions is determined by MRI-guided needle localization excisional biopsy. Patients with benign needle biopsy are followed for 2 years. Patients with benign primary lesions receive a follow up MRI scan 1 year after the initial scan. Patients with benign primary lesions and incidental enhancing lesions (IEL) are followed at 2 years. Patients with negative needle biopsies not yielding a specific diagnosis and who do not undergo subsequent excisional biopsy are followed yearly for 2 years.

PROJECTED ACCRUAL: A total of 1500 patients will be accrued for this study over 4.25 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Suspicious mammographic finding or palpable abnormality OR Suspicious clinical or ultrasound finding without associated benign mammographic features May have more than one suspicious lesion based on mammography or clinical exam if an index lesion is present Mammogram within 2 months prior to MRI scan and copy of films required of all patients 30 years of age and over Eligibility maintained if patient meets above criteria and has had: Breast implant Prior benign excisional or core biopsy at least 6 months prior to study Fine needle aspiration performed at any time Cancer in the contralateral breast No history of prior breast cancer in the study breast No benign excisional or core biopsy of the affected breast within the last 6 months

PATIENT CHARACTERISTICS: Age: 18 to 79 Sex: Women Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Cardiovascular: No implanted pacemaker Other: No implanted ferromagnetic device No ferromagnetic aneurysm clip No severe claustrophobia No ocular metal fragments No shrapnel injury No difficulty lying prone No poor venous access No impaired decision-making abilities Not pregnant

PRIOR CONCURRENT THERAPY: Not specified

Ages: 18 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 1998-05; Primary Completion 2000-06-30 (Actual); Study Completion 2000-06-30

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Schnall, PhD, Study Chair — Abramson Cancer Center at Penn Medicine
Locations (15):
- United States (12):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Roswell Park Cancer Institute, Buffalo, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
- University of Toronto, Toronto, Ontario, Canada
- Germany (2):
  - Universitaetskliniken Bonn, Bonn
  - Martin Luther Universitaet, Halle

REFERENCES:
- [Result] Schnall MD, Blume J, Bluemke DA, DeAngelis GA, DeBruhl N, Harms S, Heywang-Kobrunner SH, Hylton N, Kuhl CK, Pisano ED, Causer P, Schnitt SJ, Thickman D, Stelling CB, Weatherall PT, Lehman C, Gatsonis CA. Diagnostic architectural and dynamic features at breast MR imaging: multicenter study. Radiology. 2006 Jan;238(1):42-53. doi: 10.1148/radiol.2381042117. PMID 16373758
- [Result] Schnall MD, Blume J, Bluemke DA, Deangelis GA, Debruhl N, Harms S, Heywang-Kobrunner SH, Hylton N, Kuhl CK, Pisano ED, Causer P, Schnitt SJ, Smazal SF, Stelling CB, Lehman C, Weatherall PT, Gatsonis CA. MRI detection of distinct incidental cancer in women with primary breast cancer studied in IBMC 6883. J Surg Oncol. 2005 Oct 1;92(1):32-8. doi: 10.1002/jso.20381. PMID 16180227
- [Result] Bluemke DA, Gatsonis CA, Chen MH, DeAngelis GA, DeBruhl N, Harms S, Heywang-Kobrunner SH, Hylton N, Kuhl CK, Lehman C, Pisano ED, Causer P, Schnitt SJ, Smazal SF, Stelling CB, Weatherall PT, Schnall MD. Magnetic resonance imaging of the breast prior to biopsy. JAMA. 2004 Dec 8;292(22):2735-42. doi: 10.1001/jama.292.22.2735. PMID 15585733